CLINICAL TRIAL: NCT01951833
Title: Does Lung Clearance Index (LCI) Predict the Future Lung Disease Course in Patients With Cystic Fibrosis
Brief Title: Long Term Significance (Survival) of LCI in Patients With Cystic Fibrosis
Status: Withdrawn | Type: Observational
Sponsor: University Hospital St Luc, Brussels (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Poncin William, Physiotherapist, University Hospital St Luc, Brussels
Other Study IDs: LCI-01-St-Luc
Record Dates: First submitted 2013-03-14; First posted 2013-09-27 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2013-11

CONDITIONS: Cystic Fibrosis (CF)
Keywords: Lung clearance index (LCI)
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cystic fibrosis (Ecomedics vs NDD): No treatment, observational
  Interventions: Device: EasyOne Pro and Ecomedics
- Healthy (Ecomedics vs NDD): Free of respiratory symptoms for at least two weeks and will not have any chronic or recurrent chest problem.
  No treatment, observational
  Interventions: Device: EasyOne Pro and Ecomedics

INTERVENTIONS:
Device: EasyOne Pro and Ecomedics — LCI will be assessed with 2 different devices : EasyOne Pro and Ecomedics

SUMMARY:
The current dream in CF research is to discover safe drugs that correct the basic defect and prevent lung disease, allowing patients without significant lung damage to live nearly normal lives with a dramatic increase in life expectancy and without the burden of current treatment. The compound VX-770 (Ivacaftor Ò) is hoped to be the first milestone along this way. Progression of lung disease is now so gradual in many centres that sensitive indicators of early lung disease (small airways disease) are critically needed to assess the effects of such new treatments. In this context, assessment of ventilation inhomogeneity by the measurement called Lung clearance index (LCI) seems to be the most promising tool. However, to get approval by health authorities, new measures used in drug evaluation need to fulfill strict criteria. For LCI, the investigators still need to prove its long term significance: How well does the LCI measurement predict the long term lung disease course? Therefore, in this study the investigators want to measure LCI at baseline in a large patient cohort and establish how well it predicts the patients' disease course over the next 2 years.

DETAILED DESCRIPTION:
Patients with CF ( 6 years and older and FEV1 above 40% predicted) will be invited to participate in this prospective non interventional study in 2 CF centers ( UCL and UZ Leuven). Jointly we take care of more than 40 % of the Belgian CF population. Median FEV1 of children (6 - <18 y, n >120) from these CTN centers is high ( around 100% pred), defining a study group of great interest in the current context.

To assess the predictive value of LCI over 2 years, the time to next pulmonary exacerbation will be evaluated in the entire cohort. To assess the predictive value of LCI over 2 years, the time to next pulmonary exacerbation will be evaluated in the entire cohort.

Repeat LCI measurements will be done at subsequent patient visits.

2 devices measuring the LCI will be tested and compared : Ecomedics and NDD.

LCI and spirometry will be measured in 120 healthy Belgian children and young adults. These subjects must be free of respiratory symptoms for at least two weeks and will not have any chronic or recurrent chest problem.

ELIGIBILITY:
Inclusion Criteria:

* FEV1(% predicted) > 40%

Exclusion Criteria:

* FEV1(% predicted) < 40%
* Exacerbation during baseline measurement

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Cystic Fibrosis ( 6 years and older and FEV1 above 40% predicted) will be invited to participate in this prospective non interventional study in 2 CF centers (UCL and UZ Leuven)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Lung Clearance Index (Predictive value and change of) | Baseline, 1 week, 3 months and 2 years
  Evaluation of LCI is repeated at 1 week and 3 months to assess short and intermediate repeatability.
  LCI and spirometry will be repeated after 22-24 months after the baseline measurement. This will allow to evaluate tracking of LCI as well as FEV1 % predicted in the total patient cohort as well as in the patients with FEV1 above 80% predicted.

SECONDARY OUTCOMES:
FEV1 (Predictive value and change of) | baseline and 2 years
  LCI and spirometry will be repeated after 22-24 months after the baseline measurement. This will allow to evaluate tracking of LCI as well as FEV1 % predicted in the total patient cohort as well as in the patients with FEV1 above 80% predicted.

OTHER OUTCOMES:
Symptom score | 1 week, 3 months
  Symptom score is calculated at 1 week and 3 months to ensure a stable disease of the patient to avoid bias during the calculation of LCI repeatability.

CONTACTS AND LOCATIONS:
Overall Officials: Lebecque Patrick, PhD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Poncin William, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc (UCL), Woluwé-Saint-Lambert, Brussels Capital, Belgium